CLINICAL TRIAL: NCT02898012
Title: Temozolomide Plus Bevacizumab Chemotherapy in Supratentorial Glioblastoma in 70 Years and Older Patients With an Impaired Functional Status (KPS<70)
Brief Title: Temozolomide Plus Bevacizumab in Supratentorial Glioblastoma in 70 Years and Older Patients With an Impaired Functional Status
Acronym: ATAG
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P081213
Record Dates: First submitted 2016-07-31; First posted 2016-09-13 (Estimated); Last update posted 2016-09-13 (Estimated); Status verified 2016-07

CONDITIONS: Glioblastoma Multiforme; Primary Brain Tumor
Keywords: Glioblastoma Multiforme; temozolomide; bevacizumab
MeSH Terms: conditions — Glioblastoma; Brain Neoplasms | interventions — Temozolomide; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Temozolomide and Bevacizumab (Experimental): Single experimental arm with two drugs : Temozolomide and Bevacizumab
  Interventions: Drug: Temozolomide; Drug: Bevacizumab

INTERVENTIONS:
Drug: Temozolomide — Temozolomide (TMZ) Temozolomide (TMZ) administered at 130-150 mg/m2 for 5 consecutive days every 4 weeks up to 12 cycles. IV or oral administration was allowed according to the clinical status. TMZ starts at 130 mgs/m2 and increase to 150 mgs/m2 during the second cycle in the absence of hematologic toxicity. In the case of grade 3 or 4 toxicity, the dose for the next cycle is decreased to 110 mg/m2. If the grade 3 or 4 toxicity persists at a dose of 110 mg/m2, treatment is discontinued.
Drug: Bevacizumab — Bevacizumab (Bev) administered at a dose of 10 mgs/kg every 2 weeks. Bev was interrupted in cases of wound healing disturbances, gastrointestinal perforation, intestinal occlusion, fistula, uncontrolled hypertension, nephrotic syndrome, grade 4 or recurrent grade 3 thromboembolic events, arterial thrombosis, hemorrhage > grade 2, left ventricular failure, or posterior reversible leukoencephalopathy.

SUMMARY:
The optimal treatment of glioblastoma multiforme (GBM) in patients aged ≥70 years with a Karnofsky performance status (KPS) <70 is unestablished. This clinical trial evaluated the efficacy and safety of upfront temozolomide (TMZ) and bevacizumab (Bev) in patients aged ≥70 years and a KPS <70.

DETAILED DESCRIPTION:
Elderly patients aged 65 years and older account for approximately 45% of GBM patients, and this figure is expected to rise concurrently with the aging population of most countries. Unfortunately, few trials have been performed in this setting. In elderly patients with good functional status (KPS >70), radiotherapy (RT) prolongs overall survival (OS) without causing a detriment in quality of life compared with palliative care alone. Recently, it was shown that TMZ could be an alternative to RT. In elderly patients with poor functional status at symptom onset (KPS < 70), RT does not appear to be a satisfactory option in this frail population; however, investigators previously found that TMZ alone was associated with improvements in functional status in 1/3 of cases and appeared to increase survival compared with supportive care alone, especially in methylated MGMT promoter patients.

Bevacizumab (Bev) is an antiangiogenic monoclonal antibody targeting VEGF (vascular endothelial growth factor) that is currently used in recurrent GBM, particularly in combination with alkylating agents. Its effect as first line treatment in combination with TMZ and RT is controversial.

In this study, investigators evaluated the efficacy and safety of the upfront combination of TMZ + Bev as an initial treatment for elderly patients with GBM and impaired functional status (KPS <70).

ELIGIBILITY:
Inclusion Criteria:

* Supratentorial Glioblastoma diagnosed by biopsy.
* Patients aged ≥ 70 years
* KPS >30 and < 70
* Life expectancy > or = 8 weeks
* Patients were enrolled at least 14 days after stereotactic biopsy and 28 days after surgical biopsy.
* CT or brain MRI was performed within 4 weeks before treatment to rule out haemorrhage.
* Included to health social security system
* Medical assessment previous to inclusion
* Informed consent form

Exclusion Criteria:

* Previous treatment with Surgical resection, RT or chemotherapy to the tumor.
* Hemoglobin level < 9 g%
* Absolute neutrophil count < 1500
* Platelet count < 100.000
* ASAT or ALAT levels more than 3 times the upper limit of normal.
* Bilirubin levels more than 2 times the upper limit of normal
* Creatinin more than 1.5 times the upper limit of normal
* Untreated high blood pressure >150/100 mmHg
* Congestive cardiac failure
* Proteinuria > 1 gr/24h
* INR > 1.5 the upper limit of normal
* Recent symptomatic haemorrhage
* History of abnormal wound healing
* Gastrointestinal fistula
* Haemoptysis > grade 2 (NCI-CTC)
* Intracranial abscess
* Coagulation disorder
* Active infection requiring intravenous antibiotics
* Vascular disease (including myocardial infarction, unstable angina, cerebrovascular disease, peripheral arterial or aortic disease) in the previous 6 months
* Malignancy diagnosed in the previous 5 years (except basocellular skin cancer and in situ cervix cancer)
* Allergy to dacarbazine, Bevacizumab, Temozolomide or their excipients, recombinant human monoclonal antibodies, or ovarian cells of Chinese hamsters.

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-10; Primary Completion 2013-05 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Median Overall Survival (OS) | OS calculated from the date of surgery until death or up to 36 months.
  OS calculated from the date of surgery until death from any cause or up to 36 months.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | PFS calculated from the date of surgery until the date of first documented progression or up to 36 months.
  PFS calculated from the date of surgery to the date of progression or death or up to 36 months.
Toxicity grade according to the National Cancer Institute Common Toxicity Criteria (NCI CTCAE, version 3.0) | Assessment every 2 weeks until 12 months
  Assessment every 2 weeks until 12 months by physical and neurological examinations, complete blood counts and urine strip tests. Toxicity was graded according to the National Cancer Institute Common Toxicity Criteria (NCI CTCAE, version 3.0).
Health-related quality of life using QLQ-C30 questionnaire | at baseline and every month until 12 months
  The QLQ-C30 questionnaire includes 30 questions comprising five functioning scales (physical, role, emotional, cognitive and social), three symptom scales (fatigue, vomiting and pain) and six single item scales (dyspnea, insomnia, constipation, anorexia, diarrhea, and financial difficulties).
Health-related quality of life using QLQ-BN20 | at baseline and every month until 12 months
  The QLQ-BN20 questionnaire includes 20 items covering functional deficits, symptoms, toxic effects of treatment, and uncertainty about the future.
Cognitive assessment MMSEs | at baseline and they were repeated every month until 12 months
  The MMSE was used as a measure of general cognitive status. Higher scores on this exam, which uses a 30-point scale, indicate better cognitive function.
Radiological responses | Neuroimaging evaluation repeated every 2 months until 12 months
  Response assessment in neuro-oncology (RANO) criteria

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Yves Delattre, MD-PhD, Principal Investigator — Pôle MSN, Groupe Hospitalier Pitié-Salpêtrière
Locations (1):
- Groupe Hospitalier Pitié-Salpêtrière, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dolecek TA, Propp JM, Stroup NE, Kruchko C. CBTRUS statistical report: primary brain and central nervous system tumors diagnosed in the United States in 2005-2009. Neuro Oncol. 2012 Nov;14 Suppl 5(Suppl 5):v1-49. doi: 10.1093/neuonc/nos218. No abstract available. PMID 23095881
- [Background] Fleury A, Menegoz F, Grosclaude P, Daures JP, Henry-Amar M, Raverdy N, Schaffer P, Poisson M, Delattre JY. Descriptive epidemiology of cerebral gliomas in France. Cancer. 1997 Mar 15;79(6):1195-202. doi: 10.1002/(sici)1097-0142(19970315)79:63.0.co;2-v. PMID 9070498
- [Background] Keime-Guibert F, Chinot O, Taillandier L, Cartalat-Carel S, Frenay M, Kantor G, Guillamo JS, Jadaud E, Colin P, Bondiau PY, Menei P, Loiseau H, Bernier V, Honnorat J, Barrie M, Mokhtari K, Mazeron JJ, Bissery A, Delattre JY; Association of French-Speaking Neuro-Oncologists. Radiotherapy for glioblastoma in the elderly. N Engl J Med. 2007 Apr 12;356(15):1527-35. doi: 10.1056/NEJMoa065901. PMID 17429084
- [Background] Malmstrom A, Gronberg BH, Marosi C, Stupp R, Frappaz D, Schultz H, Abacioglu U, Tavelin B, Lhermitte B, Hegi ME, Rosell J, Henriksson R; Nordic Clinical Brain Tumour Study Group (NCBTSG). Temozolomide versus standard 6-week radiotherapy versus hypofractionated radiotherapy in patients older than 60 years with glioblastoma: the Nordic randomised, phase 3 trial. Lancet Oncol. 2012 Sep;13(9):916-26. doi: 10.1016/S1470-2045(12)70265-6. Epub 2012 Aug 8. PMID 22877848
- [Background] Wick W, Platten M, Meisner C, Felsberg J, Tabatabai G, Simon M, Nikkhah G, Papsdorf K, Steinbach JP, Sabel M, Combs SE, Vesper J, Braun C, Meixensberger J, Ketter R, Mayer-Steinacker R, Reifenberger G, Weller M; NOA-08 Study Group of Neuro-oncology Working Group (NOA) of German Cancer Society. Temozolomide chemotherapy alone versus radiotherapy alone for malignant astrocytoma in the elderly: the NOA-08 randomised, phase 3 trial. Lancet Oncol. 2012 Jul;13(7):707-15. doi: 10.1016/S1470-2045(12)70164-X. Epub 2012 May 10. PMID 22578793
- [Background] Gallego Perez-Larraya J, Ducray F, Chinot O, Catry-Thomas I, Taillandier L, Guillamo JS, Campello C, Monjour A, Cartalat-Carel S, Barrie M, Huchet A, Beauchesne P, Matta M, Mokhtari K, Tanguy ML, Honnorat J, Delattre JY. Temozolomide in elderly patients with newly diagnosed glioblastoma and poor performance status: an ANOCEF phase II trial. J Clin Oncol. 2011 Aug 1;29(22):3050-5. doi: 10.1200/JCO.2011.34.8086. Epub 2011 Jun 27. PMID 21709196
- [Background] Taal W, Oosterkamp HM, Walenkamp AM, Dubbink HJ, Beerepoot LV, Hanse MC, Buter J, Honkoop AH, Boerman D, de Vos FY, Dinjens WN, Enting RH, Taphoorn MJ, van den Berkmortel FW, Jansen RL, Brandsma D, Bromberg JE, van Heuvel I, Vernhout RM, van der Holt B, van den Bent MJ. Single-agent bevacizumab or lomustine versus a combination of bevacizumab plus lomustine in patients with recurrent glioblastoma (BELOB trial): a randomised controlled phase 2 trial. Lancet Oncol. 2014 Aug;15(9):943-53. doi: 10.1016/S1470-2045(14)70314-6. Epub 2014 Jul 15. PMID 25035291
- [Background] Stupp R, Mason WP, van den Bent MJ, Weller M, Fisher B, Taphoorn MJ, Belanger K, Brandes AA, Marosi C, Bogdahn U, Curschmann J, Janzer RC, Ludwin SK, Gorlia T, Allgeier A, Lacombe D, Cairncross JG, Eisenhauer E, Mirimanoff RO; European Organisation for Research and Treatment of Cancer Brain Tumor and Radiotherapy Groups; National Cancer Institute of Canada Clinical Trials Group. Radiotherapy plus concomitant and adjuvant temozolomide for glioblastoma. N Engl J Med. 2005 Mar 10;352(10):987-96. doi: 10.1056/NEJMoa043330. PMID 15758009
- [Background] Lou E, Peters KB, Sumrall AL, Desjardins A, Reardon DA, Lipp ES, Herndon JE 2nd, Coan A, Bailey L, Turner S, Friedman HS, Vredenburgh JJ. Phase II trial of upfront bevacizumab and temozolomide for unresectable or multifocal glioblastoma. Cancer Med. 2013 Apr;2(2):185-95. doi: 10.1002/cam4.58. Epub 2013 Jan 24. PMID 23634286
- [Background] Friedman HS, Prados MD, Wen PY, Mikkelsen T, Schiff D, Abrey LE, Yung WK, Paleologos N, Nicholas MK, Jensen R, Vredenburgh J, Huang J, Zheng M, Cloughesy T. Bevacizumab alone and in combination with irinotecan in recurrent glioblastoma. J Clin Oncol. 2009 Oct 1;27(28):4733-40. doi: 10.1200/JCO.2008.19.8721. Epub 2009 Aug 31. PMID 19720927
- [Background] Scott JG, Bauchet L, Fraum TJ, Nayak L, Cooper AR, Chao ST, Suh JH, Vogelbaum MA, Peereboom DM, Zouaoui S, Mathieu-Daude H, Fabbro-Peray P, Rigau V, Taillandier L, Abrey LE, DeAngelis LM, Shih JH, Iwamoto FM. Recursive partitioning analysis of prognostic factors for glioblastoma patients aged 70 years or older. Cancer. 2012 Nov 15;118(22):5595-600. doi: 10.1002/cncr.27570. Epub 2012 Apr 19. PMID 22517216
- [Background] Rosati G, Avallone A, Aprile G, Butera A, Reggiardo G, Bilancia D. XELOX and bevacizumab followed by single-agent bevacizumab as maintenance therapy as first-line treatment in elderly patients with advanced colorectal cancer: the boxe study. Cancer Chemother Pharmacol. 2013 Jan;71(1):257-64. doi: 10.1007/s00280-012-2004-x. Epub 2012 Oct 26. PMID 23100174
- [Background] Cunningham D, Lang I, Marcuello E, Lorusso V, Ocvirk J, Shin DB, Jonker D, Osborne S, Andre N, Waterkamp D, Saunders MP; AVEX study investigators. Bevacizumab plus capecitabine versus capecitabine alone in elderly patients with previously untreated metastatic colorectal cancer (AVEX): an open-label, randomised phase 3 trial. Lancet Oncol. 2013 Oct;14(11):1077-1085. doi: 10.1016/S1470-2045(13)70154-2. Epub 2013 Sep 10. PMID 24028813
- [Background] Biganzoli L, Di Vincenzo E, Jiang Z, Lichinitser M, Shen Z, Delva R, Bogdanova N, Vivanco GL, Chen Z, Cheng Y, Just M, Espie M, Vinholes J, Hamm C, Crivellari D, Chmielowska E, Semiglazov V, Dalenc F, Smith I. First-line bevacizumab-containing therapy for breast cancer: results in patients aged>/=70 years treated in the ATHENA study. Ann Oncol. 2012 Jan;23(1):111-118. doi: 10.1093/annonc/mdr043. Epub 2011 Mar 28. PMID 21444356
- [Background] Laskin J, Crino L, Felip E, Franke F, Gorbunova V, Groen H, Jiang GL, Reck M, Schneider CP. Safety and efficacy of first-line bevacizumab plus chemotherapy in elderly patients with advanced or recurrent nonsquamous non-small cell lung cancer: safety of avastin in lung trial (MO19390). J Thorac Oncol. 2012 Jan;7(1):203-11. doi: 10.1097/JTO.0b013e3182370e02. PMID 22173662
- [Background] Chauffert B, Feuvret L, Bonnetain F, Taillandier L, Frappaz D, Taillia H, Schott R, Honnorat J, Fabbro M, Tennevet I, Ghiringhelli F, Guillamo JS, Durando X, Castera D, Frenay M, Campello C, Dalban C, Skrzypski J, Chinot O. Randomized phase II trial of irinotecan and bevacizumab as neo-adjuvant and adjuvant to temozolomide-based chemoradiation compared with temozolomide-chemoradiation for unresectable glioblastoma: final results of the TEMAVIR study from ANOCEFdagger. Ann Oncol. 2014 Jul;25(7):1442-1447. doi: 10.1093/annonc/mdu148. Epub 2014 Apr 9. PMID 24723487
- [Background] Chinot OL, Wick W, Mason W, Henriksson R, Saran F, Nishikawa R, Carpentier AF, Hoang-Xuan K, Kavan P, Cernea D, Brandes AA, Hilton M, Abrey L, Cloughesy T. Bevacizumab plus radiotherapy-temozolomide for newly diagnosed glioblastoma. N Engl J Med. 2014 Feb 20;370(8):709-22. doi: 10.1056/NEJMoa1308345. PMID 24552318
- [Background] Gilbert MR, Dignam JJ, Armstrong TS, Wefel JS, Blumenthal DT, Vogelbaum MA, Colman H, Chakravarti A, Pugh S, Won M, Jeraj R, Brown PD, Jaeckle KA, Schiff D, Stieber VW, Brachman DG, Werner-Wasik M, Tremont-Lukats IW, Sulman EP, Aldape KD, Curran WJ Jr, Mehta MP. A randomized trial of bevacizumab for newly diagnosed glioblastoma. N Engl J Med. 2014 Feb 20;370(8):699-708. doi: 10.1056/NEJMoa1308573. PMID 24552317
- [Background] Fardet L, Feve B. Systemic glucocorticoid therapy: a review of its metabolic and cardiovascular adverse events. Drugs. 2014 Oct;74(15):1731-45. doi: 10.1007/s40265-014-0282-9. PMID 25204470
- [Derived] Reyes-Botero G, Cartalat-Carel S, Chinot OL, Barrie M, Taillandier L, Beauchesne P, Catry-Thomas I, Barriere J, Guillamo JS, Fabbro M, Frappaz D, Benouaich-Amiel A, Le Rhun E, Campello C, Tennevet I, Ghiringhelli F, Tanguy ML, Mokhtari K, Honnorat J, Delattre JY. Temozolomide Plus Bevacizumab in Elderly Patients with Newly Diagnosed Glioblastoma and Poor Performance Status: An ANOCEF Phase II Trial (ATAG). Oncologist. 2018 May;23(5):524-e44. doi: 10.1634/theoncologist.2017-0689. Epub 2018 Feb 22. PMID 29472310